CLINICAL TRIAL: NCT01028820
Title: Pilot Study of the Effect of Aripiprazole Treatment in Autism Spectrum Disorders on Functional Magnetic Resonance Imaging (fMRI) Activation Patterns and Symptoms
Brief Title: FMRI Brain Activation of Aripiprazole Treatment in Autism Spectrum Disorders
Acronym: AripfMRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090795; K23MH081285 (NIH)
Record Dates: First submitted 2009-12-04; First posted 2009-12-09 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; asperger's; repetitive; restricted; compulsions
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Compulsive Behavior | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label, Flexible-Dose Aripiprazole (Experimental): This is a single group assignment pharmacodynamics study in which all study participants are given an open-label, flexible dose of aripiprazole for up to 8 weeks.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 8 weeks, starting dosage 5mg titrating up 5mg every week as needed to maximum dosage of 25mg daily
  Other Names: Abilify

SUMMARY:
This is an 8 week research study of aripiprazole (abilify) which is used to reduce irritable behaviors in autism spectrum disorders. All participants will receive active study medication. Participants will also receive diagnostic and cognitive evaluations at no cost. Participants will be required to undergo two fMRI (functional magnetic resonance imaging scans) where we will take pictures of your brain while performing simple tasks.

ELIGIBILITY:
Inclusion Criteria:

* male or female of any race or ethnicity
* ambulatory status (outpatient) at time of consent
* age 10-55 inclusive at time of consent
* clinical diagnosis of autism spectrum disorder and meets screening criteria on the Social Communication Questionnaire as well as either the Autism Diagnostic Observation Schedule (ADOS) or the Autism Diagnostic Interview-Revised (ADI-R) administered by raters trained to research reliability.
* estimated IQ greater than 70 and capable of making an informed decision based on assessment of their understanding and judgment
* Children's Yale-Brown Obsessive Compulsive Scale: Modified for Pervasive Developmental Disorders (PDD-CYBOCS) > 8 as assessed during telephone screening.
* Free of psychoactive medication for at least: one month for fluoxetine; two weeks for other SSRIs and neuroleptics; and five days for stimulants prior to MRI scanning [excepting stable doses (greater than three months duration) of anticonvulsant medication for seizure disorder]
* Currently taking psychoactive medication that is not providing sufficient relief of repetitive behaviors and willing to discontinue all psychoactive medication for the duration of the study.
* Judged reliable for medication compliance and agreeing to keep follow-up study appointments.

Exclusion Criteria:

* Age less than 10 years or greater than 55 years at time of consent
* Estimated IQ less than 70
* Uncontrolled epilepsy (seizure within 6 months prior to consent)
* Presence of medical conditions that might interfere with participation, or where participation would be contraindicated.
* History of neurological injury: head trauma, poorly-controlled seizure disorder (seizure within the preceding six months), stroke, prior neurosurgery, or under the care of a neurologist or neurosurgeon as determined by interview
* History of claustrophobia
* Implanted or irremovable metal in the body (including certain tattoos and permanent make-up).
* Current pregnancy in females
* Inability to communicate satisfactorily and directly (without a translator) in English
* Medical contraindications to aripiprazole therapy as determined by history (including induction of neuroleptic malignant syndrome, dystonic reaction, or known drug allergy)
* Ongoing need for psychoactive medication other than study medication [excepting stable doses (greater than 3 months duration) of anticonvulsant medication for seizure disorder or diphenhydramine for sleep
* prior history of aripiprazole treatment failure at appropriate doses and duration
* clinically significant low white blood cell count at baseline

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina; Gabriel Dichter, PhD, Principal Investigator — University of North Carolina and Duke University; Cheryl O Alderman, BS, Study Director — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We planned to recruit participants through the NDRC Registry and Division TEACCH, as well as utilizing radio and television ads on various stations. We also posted brochures and flyers in public locations and attended conferences in order to hand out study-specific information. 13 subjects began the study and only one of those failed to complete.
Pre-assignment Details: In order to participate in the research study, subjects must have been washed out from psychoactive medication for at least one month for fluoxetine, two weeks for other SSRIs and neuroleptics and five days for stimulants prior to MRI scanning, with the exception of stable doses greater than three months duration of medication for seizure disorder.
Groups:
- Open-Label, Flexible-Dose Aripiprazole: This is a single group assignment pharmacodynamics study in which all study participants are given an open-label, flexible dose of aripiprazole for up to 8 weeks.
  Aripiprazole : 8 weeks, starting dosage 5mg titrating up 5mg every week as needed to maximum dosage of 25mg daily
Period: Overall Study
Arm/Group | Open-Label, Flexible-Dose Aripiprazole
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label, Flexible-Dose Aripiprazole
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.31 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Total Repetitive Behavior Scale - Revised (RBS_R)
Description: The RBS-R is an assessment that includes Sameness, Self-Injurious Behavior, Ritualistic, Compulsive, and Restrictive Behavior subscales. The assessments are completed by caregivers for the past week, with consideration of frequency,ease of redirecting and extent to which behavior interferes with functioning compared to a typically developing child of the same age and gender. Scores are rated from 0 - behavior does not occur to 3 - behavior occurs and is a serious problem. There are 43 items and 5 subscales. Higher scores indicate greater symptom severity. total score is the sum of all items in all subscales.
  The subscales are stereotyped behaviors 6 items, self-injurious behaviors 8 items, Compulsive behaviors- 8 items, Ritualistic Behaviors 6 items, Sameness 11 items, restricted behaviors 4 items.Total score ranges from 0 to 129.
Time Frame: baseline week 0, 8 weeks
Population: All randomized participants' scores were analyzed using the RBS-R measure. Higher values reflect worse outcomes (greater symptom severity). Subscales are added to compute the total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open-Label, Flexible-Dose Aripiprazole: Baseline (Pre-Dose); Open-Label, Flexible-Dose Aripiprazole: 8 Weeks (Post-Dose): This is a single group assignment pharmacodynamics study in which all study participants are given an open-label, flexible dose of aripiprazole for up to 8 weeks.
  Aripiprazole : 8 weeks, starting dosage 5mg titrating up 5mg every week as needed to maximum dosage of 25mg daily
Arm/Group | Open-Label, Flexible-Dose Aripiprazole: Baseline (Pre-Dose) | Open-Label, Flexible-Dose Aripiprazole: 8 Weeks (Post-Dose)
Number analyzed (Participants) | 13 | 13
units on a scale | 42.2 (18.37) | 20.5 (13.79)

2. Primary Outcome: Baseline and Week 8scores on Children's Yale-Brown Obsessive Compulsive Scale - Pervasive Developmental Disorder Version
Description: The Children's Yale-Brown Obsessive Compulsive Scale - Pervasive Developmental Disorder Version (CY-BOCS-PDD) is a clinician-rated interview designed to evaluate repetitive behavior in children with pervasive developmental disorders (PDDs). It is a modification of the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS), developed to assess typically-developing children with obsessive compulsive behavior. Because of language limitations in children with PDDs the CY-BOCS-PDD only includes the five compulsion items: Time Spent, Interference, Distress, Resistance of repetitive behavior, and Control of repetitive behavior. Each item is rated from 0 (none) through 4 (extreme), and scores can range from 0 to 20, with higher scores reflecting more severe symptoms. Usually a score > than 8 is considered clinically significant.
Time Frame: Baseline ("Pre-Dose") to 8 Weeks ("Post-Dose")
Population: All randomized participants' scores were analyzed using the PDD-CYBOCS measure. Higher values reflect worse outcomes. Subscales are added to compute the total score (total score does not include compulsion free-interval and peculiarity of the behavior.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Open-Label, Flexible-Dose Aripiprazole: Baseline (Pre-Dose) | Open-Label, Flexible-Dose Aripiprazole: 8 Weeks (Post-Dose)
Number analyzed (Participants) | 13 | 13
Scores on a scale | 12.7 (2.250) | 8.6 (3.50)

ADVERSE EVENTS:
Arm/Group | Open-Label, Flexible-Dose Aripiprazole
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label, Flexible-Dose Aripiprazole (N=13)
Anxiety (Social circumstances) | 2 (2)
Body Pain (General disorders) | 3 (3)
Depressed Mood (Psychiatric disorders) | 1 (1)
Drowsiness (General disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Increased Appetite (Metabolism and nutrition disorders) | 3 (3)
Increased Sleep (General disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Restlessness (General disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremors (Nervous system disorders) | 1 (1)
Urination (Renal and urinary disorders) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The present study had 13 subjects. Due to sample size, analysis reflected an exploratory approach. If a mechanism for predicting RRB improvement is found in a study with a larger N, we could better understand therapies targeting core symptoms of ASD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No